CLINICAL TRIAL: NCT05751434
Title: Phase 2 Trial of Exercise Therapy on Markers of Progression in Localized Prostate Cancer
Brief Title: A Study on the Effects of Exercise Therapy on Signs of Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-419
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Localized Prostate Carcinoma
Keywords: Prostate Cancer; Prostate Adenocarcinoma; Localized Prostate Carcinoma; exercise therapy; Memorial Sloan Kettering Cancer Center; 22-419
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants Assigned to Exercise Therapy (Experimental): Participants with histologically confirmed localized prostate cancer undergoing active surveillance
  Interventions: Behavioral: Exercise Therapy
- Participants Assigned to Usual Care (No Intervention): Participants with histologically confirmed localized prostate cancer undergoing active surveillance

INTERVENTIONS:
Behavioral: Exercise Therapy — The intervention will consist of exercise therapy, individualized, walking delivered following a non-linear (i.e., exercise dose is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule, up to 5 individual treatment sessions/week to achieve a cumulative total duration of 225 to 300 mins/wk until the participant's next standard of care prostate biopsy (about 6-12 months).
  Arms: Participants Assigned to Exercise Therapy

SUMMARY:
The purpose of this study is to find out the effects of exercise therapy on indicators of prostate cancer in people with low-risk prostate cancer who are on active surveillance. The exercise therapy in this study will be regular home-based walking sessions on a treadmill, and that therapy will be assigned by an exercise physiologist (a medical professional who studies how exercise affects the human body). Some participants in this study will have the assigned exercise therapy, and some participants will participate in their usual exercise routines. Researchers will compare how the assigned exercise therapy and the usual exercise routines affect indicators of prostate cancer in participants. This study will not provide treatment for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Men with histologically confirmed localized prostate cancer undergoing active surveillance.
* Inactive, defined as not meeting the national exercise guidelines for cancer patients (<150 minutes/week of moderate or vigorous exercise)43 as assessed by remote activity and heart rate tracking for a 7-day period prior to study entry (general physical activity screening assessment via smart watch).
* Screening clearance by an MSK Exercise Physiologist (i.e., review of ECG)
* BMI <40 kg/m^2
* Cleared for exercise participation as per pre-screening clearance via the Physical Activity Readiness Questionnaire (PAR-Q+) (Appendix B)

Exclusion Criteria:

* Enrollment in any other program that may alter the impact of exercise on tumor outcomes (e.g., weight loss program)
* Any neoadjuvant anticancer treatment of any kind for prostate cancer in the last 5 years
* Any history of systemic anticancer therapy in the last 15 years
* Distant metastatic malignancy of any kind
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in molecular, radiologic, and pathologic nimbosus hallmarks from baseline to follow-up | 6-12 months
  The phenomenon of multiple independent prognostic features that moderately correlate with one another has been termed Nimbosus, "a gathering of storm clouds". The more Nimbosus hallmarks present in a tumor, the more aggressive it is likely to be, and the greater the chance that it will escape the prostate leading to nodal and distal metastatic spread. Nimbosus hallmarks provides a targetable set of biomarkers to test in a RCT of exercise therapy in localized prostate cancer.
  Molecular end points will be evaluated on FFPE tumor samples obtained from a total of two ultrasound-guided transrectal prostate biopsies performed at pretreatment (diagnostic biopsy) and post-intervention around month 6-12 (confirmatory biopsy), as per standard procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of California, Los Angeles (Data and Specimen Analysis Only), Los Angeles, California
  - Hartford Healthcare Alliance (Data collection only), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org